CLINICAL TRIAL: NCT06280053
Title: The Clinical Safety and Effectiveness of HealiAid Collagen Wound Dressing in the Treatment of Different Wounds
Brief Title: HealiAid in the Treatment of Different Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maxigen Biotech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 103-3024A3
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Venous Ulcers; Bedsores; Diabetic Foot Wound; Burn Wound
Keywords: Collagen Wound Dressing; Post-marketing Study
MeSH Terms: conditions — Varicose Ulcer; Pressure Ulcer; Burns

STUDY DESIGN:
Intervention Model Description: The patients' wound conditions were divided into four types: venous ulcers, bedsores, diabetic foot wounds and burn wounds.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HealiAid group (Experimental): The patients' wound conditions were divided into three types: venous ulcers, bedsores and burn wounds.
  Interventions: Device: HealiAid Collagen Wound Dressing

INTERVENTIONS:
Device: HealiAid Collagen Wound Dressing — HealiAid is an absorbable collagen wound dressing. It is fabricated by fibrous collagen matrix, in which the collagen is purified from bovine Achilles tendons. HealiAid can be applied easily by covering directly to the clean wound sites.

SUMMARY:
The goal of this open-label, post-market clinical follow-up study is to demonstrate the safety and effectiveness of HealiAid Collagen Wound Dressing in patients classified into different types of wounds: venous ulcers, bedsores, diabetic foot wounds and burn wounds.

The main questions it aims to answer are:

1. The wound healing which was defined as the percentage of area change.
2. The duration of wound healing.
3. The granulation tissue growth of the wound.
4. The wound exudate.
5. Safety Indicators of which incidences after treatment.

HealiAid will be applied to eligible subjects who will later be followed up for 12 weeks.

DETAILED DESCRIPTION:
An open-label study will be performed in single center to monitor about 6 patients in each types of wounds: venous ulcers, bedsores, diabetic foot wounds and burn wounds, totally 24 patients, after the treatment of using HealiAid Collagen Wound Dressing (MAXIGEN BIOTECH INC., Taiwan) directly on the wound sites.

Follow-up visits will be at 1, 2, 4, 8 and 12(if needed) weeks after the treatment.

The primary endpoint of this study was the area percentage of healed wound at the 8-week post-treatment interval, which is also considered as the healing condition of the wound.

The secondary endpoints of this study were included the duration of wound healing, granulation tissue growth, wound exudate, and the incidence of safety events.

T-test or Wilcoxon rank-sum test will be used to test for the differences between baseline and each visit. Statistical significance was established at p < 0.05.

The actual enrollment of this study was 6 participants each in the venous ulcers, bedsores, and burn wounds, while no patients with diabetic foot wounds were recruited, resulting in a total of 18 participants.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age with wounds.
* The venous ulcer has been present for at least 30 days without healing, graded as stage 3, and the wound is at least 1 cm^2 (maximum length x maximum width).
* Diabetic foot wound is classified as Wagner grade 2, and the wound is at least 1cm^2 (maximum length × maximum width).
* Bedsore (NPUAP) is graded as level 2, and the wound is at least 1cm^2 (Maximum length × maximum width).
* Burn wound is classified as grade 2, and the wound is at least 1cm^2 (maximum length × maximum width).
* The limbs of patients with venous ulcers and diabetes are assessed using Doppler to measure blood circulation, confirming adequate blood flow in the affected tissues.
* After a complete debridement operation, confirm that there is no necrotic or viable lesion tissue.

Exclusion Criteria:

* There is an inflammatory response clinically.
* A wound site with bone exposure.
* Existing conditions or diseases may affect wound healing(e.g., cancer, vasculitis, connective tissue disorders, or any immune system disorders).
* Alcohol abuse.
* Within the past 30 days prior to enrollment, any use of medications that may affect wound healing, such as those associated with dialysis, steroids, immunosuppressants, radiation therapy, or chemotherapy.
* There are multiple ulcer wounds present on the same limb affected by the lesion.
* Pregnant or lactating women.
* It is known that there has been a previous allergic reaction to any component of the dressing.
* Allergic to collagen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-03-02 (Actual); Primary Completion 2018-04-11 (Actual); Study Completion 2018-10-26 (Actual)

PRIMARY OUTCOMES:
Wound Healing | Baseline, 8 weeks after treatment
  The wound healing was defined as the percentage of area change at baseline and 8 weeks after treatment.
  The wound area was calculated by multiplying the length (direction from head to leg) by the width (widest part of the wound site, perpendicular to the length).
  The percentage of area change was calculated by the formula: (baseline wound area minus 8-week wound area)/baseline wound area *100%.

SECONDARY OUTCOMES:
Wound Healing | Baseline, 1, 2, 4, 12(if needed) weeks after treatment
  The wound healing was defined as the percentage of area change at baseline and 1, 2, 4 weeks after treatment.
  The wound area was calculated by multiplying the length (direction from head to leg) by the width (widest part of the wound site, perpendicular to the length).
  The percentage of area change was calculated by the formula: (baseline wound area minus 1, 2 or 4-week wound area)/baseline wound area *100%.
Duration of Wound Healing | Baseline, 1, 2, 4, 12(if needed) weeks after treatment
  The duration of wound healing was recorded using the subjects' diaries, which indicated the time when the wound completely healed.
Granulation Tissue Growth | Baseline, 1, 2, 4, 8, 12(if needed) weeks after treatment
  The granulation tissue growth was defined using a scale of 6 grades.
  * 0: the wound site is either completely healed or shallow.
  * 1: the granulation tissue occupied 90% of wound area
  * 2: the granulation tissue occupied ≥50%, <90% of wound area
  * 3: the granulation tissue occupied ≥10%, <50% of wound area
  * 4: the granulation tissue occupied <10% of wound area
  * 5: No granulation tissue present
Wound Exudate | Baseline, 1, 2, 4, 8, 12(if needed) weeks after treatment
  The extent of wound exudate was classified as 4 grades.
  * 0: No wound exudate
  * 1: Small amount of wound exudate, may not require daily dressing changes
  * 2: Moderate amount of wound exudate, requires daily dressing changes
  * 3: Large amount of wound exudate, dressing changes at least twice daily
Incidence of Safety Events | week 0 to week 12
  The safety events were defined as the wound site infection/inflammation and scoring as:
  * 0: No signs of infection or inflammation.
  * 1: Redness, swelling, heat, and pain that indicated inflammation.
  * 2: Clear signs of infection such as inflammation, purulence, or odor.
  * 3: Systemic symptoms such as fever.
  Other safety events such as allergic reaction was scored as:
  * 0: No reaction
  * 1: Doubtful reaction
  * 2: Weak reaction
  * 3: Strong reaction

CONTACTS AND LOCATIONS:
Overall Officials: Huang-Kai Kao, Doctor, Principal Investigator — Chang Gung Memorial Hospital